CLINICAL TRIAL: NCT04902300
Title: Prevalence of Internet Addiction Among Adolescent
Acronym: ADDICT-NET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-002-ADDICT-NET
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Internet Addiction
Keywords: Adolescent; Internet addiction; Prevalence
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent: adolescent attending high school
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — evaluation of internet addiction

SUMMARY:
Internet is now a tool available 24 hours a day, at a lower cost and accessible almost anywhere. Internet addiction could be defined as the inability to control one's Internet use and the continuation of this behavior despite the occurrence of negative consequences.

Adolescence is a time of vulnerability to addiction, due to social and neurobiological factors.

DETAILED DESCRIPTION:
The aim of the study is to evaluate prevalence of internet addiction among adolescent attending high school

ELIGIBILITY:
Inclusion Criteria:

* adolescent attending high school
* agreeing to participate in the study

Exclusion Criteria:

* None

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent attending high school
Sampling Method: Non-Probability Sample
Enrollment: 4750 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
internet addiction | Day 0
  Internet addiction evaluated using Compulsive Internet Use Scale (CIUS-9). CIUS-9 includes 9 items. Each item is coded from 0 to 4 points. The overall score ranges from 0 to 36 points. The higher the score, the more compulsive the internet behavior. A score greater than or equal to 18 defines an internet addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CORPEL, MD, Principal Investigator — Université de Reims Champagne-Ardenne
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France